CLINICAL TRIAL: NCT01538472
Title: Y Zevalin, BEAM and Rituximab In Autologous Stem Cell Transplantation (ASCT) For Lymphoma
Brief Title: Y Zevalin and BEAM in Autologous Stem Cell Transplantation (ASCT) for Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0123
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Lymphoma
Keywords: Lymphoma; Relapse B-cell CD20+ non-Hodgkin's lymphoma; High-dose BEAM chemotherapy; Y Zevalin; In Zevalin; Rituxan; Rituximab; BCNU; 1,3-bis(2-chloroethyl)-1-nitrosourea bis-chloronitrosourea; Carmustine; BiCNU; VP-16; Ara-C; Cytarabine; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride; Melphalan; Alkeran; G-CSF; Filgrastim; Neupogen; Stem cell infusion; Autologous stem cell transplantation
MeSH Terms: conditions — Lymphoma | interventions — ibritumomab tiuxetan; Rituximab; Carmustine; Etoposide; Cytarabine; Melphalan; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Y Zevalin + BEAM (Experimental): Rituxan 250 mg/m2 preceding imaging dose of 111In Zevalin (5 mCi); additional infusion 250 mg/m2 Rituxan followed by therapeutic dose of 0.4 mCi/kg 90Y Zevalin received one week after Rituxan/111In Zevalin infusions. One week later, chemotherapy received with BCNU (300 mg/m2, intravenously (IV) day -6) VP-16 (200 mg/m2 IV every 12 hours, days -5 to -2) cytarabine (200 mg/m2 IV every 12 hours, days -5 to -2) and melphalan (140 mg/m2 IV day -1). Autologous stem cell infused on day 0 then Rituximab 1000 mg/m2 on days +1, and +8 post transplantation.
  G-CSF 5 mg/kg given daily starting Day 0 till recovery of granulocytes of 4.0 * 109/L.
  Interventions: Drug: Y Zevalin; Drug: In Zevalin; Drug: Rituxan; Drug: BCNU; Drug: VP -16; Drug: Ara-C; Drug: Melphalan; Procedure: Stem Cell Infusion; Drug: G-CSF

INTERVENTIONS:
Drug: Y Zevalin — Starting dose: 0.4 mCi/kg by vein after Rituxan infusion on Day -14.
Drug: In Zevalin — Imaging dose: 5 mCi by vein following Rituxan infusion on Day -21.
Drug: Rituxan — 250 mg/m2 by vein on Day -21 and on Day -14.
  1000 mg/m2 by vein on Days +1 and +8.
  Other Names: Rituximab
Drug: BCNU — 300 mg/m2 by vein on Day -6.
  Other Names: Carmustine; BiCNU; 1,3-bis(2-chloroethyl)-1-nitrosourea bis-chloronitrosourea
Drug: VP -16 — 200 mg/m2 by vein every 12 hours on Days -5, -4, -3, and -2.
Drug: Ara-C — 200 mg/m2 by vein every 12 hours on Days -5, -4, -3,and -2.
  Other Names: Cytarabine; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Melphalan — 140 mg/m2 by vein on Day -1.
  Other Names: Alkeran
Procedure: Stem Cell Infusion — Autologous stem cell infusion on Day 0.
Drug: G-CSF — 5 mg/kg by vein daily starting Day 0 till recovery of granulocytes of 4.0 x 109/L.
  Other Names: Filgrastim; Neupogen

SUMMARY:
The goal of this clinical research study is to see if high-dose chemotherapy (BEAM) and rituximab, given together with the new drug 90Y Zevalin, followed by a transplant of blood or marrow stem cells is safe. Another goal is to learn if this treatment can help decrease the chances of the cancer coming back.

DETAILED DESCRIPTION:
BEAM chemotherapy is the standard treatment for lymphoma. BEAM is a combination of chemotherapy drugs (carmustine, cytarabine, etoposide, and melphalan). Rituximab is an antibody made from human and mouse proteins. It reacts with a certain molecule on the surface of lymphoma cells and helps the body's immune system destroy the lymphoma cells. 90Y Zevalin is also an antibody made from mouse proteins. However, it has a particle of radiation attached to it. 90Y Zevalin works by attaching to lymphoma cells, and the radiation particle destroys the lymphoma cell.

For this study, you will receive rituximab by vein followed by a dose of 111In Zevalin by vein (over 15 minutes). 111In Zevalin is different from the study drug (90Y Zevalin). 111In Zevalin has a different type of radioactive particle attached to it. This particle does not kill lymphoma cells, but it can be "seen" inside the body using a special camera (like an x-ray). 111In Zevalin is being used to predict how fast the study drug will travel in the body and how long the drug stays in the body. Doctors need to be able to see how much of the drug goes to the tumor and how much goes to normal organs to determine if it is safe to give 90Y Zevalin on an outpatient basis. A scan will be done as soon as 111In Zevalin is given and about 2-24 hours later. Scans will also be done 2-3 days later. If the radiation in the 111In Zevalin is not a threat to normal organs and bone marrow, you may receive 90Y Zevalin. Seven (7) days after the 111In Zevalin injection, you will receive a second dose of rituximab followed by a dose of 90Y Zevalin by vein (over 15 minutes).

Seven (7) days after the 90Y Zevalin injection, you will receive the BEAM combination of chemotherapy. You will receive carmustine (over 2 hours) on Day 1 of chemotherapy. You will receive cytarabine (over 2 hours) followed by etoposide (over 4 hours) twice a day on Days 2 through 5. On Day 6, you will receive melphalan (over 20 minutes). A catheter (small flexible tube) will be placed in a large vein in your chest so that the chemotherapy drugs can be given to you more easily. This is called a central venous catheter. All of the chemotherapy drugs will be given through the central venous catheter.

One day after finishing the chemotherapy, the stem cells that were collected earlier will be given back to you by vein over about 30 minutes. Starting on the same day, you will receive treatments with G-CSF by injection under the skin once a day. Treatment with G-CSF will continue until your blood counts reach a certain level.

You will receive rituximab by vein (over 6 to 8 hours) on the day after the transplant and again 1-week later.

Blood tests (about 1-2 tablespoons), urine tests, bone marrow collections, and x-rays will be done as needed to track the effects of the transplant. You will have transfusions of blood and platelets as needed. Blood tests (about 1 tablespoon) will be done once a day while you are in the hospital.

Blood tests (about 1-2 tablespoons), urine tests, bone marrow collections, x-rays, CT scans, and PET scans will be done every 3 months for 1 year and then every 6 months for 5 years to check on the status of the disease.

You will be asked to give some extra blood samples (around 1 tablespoon each) at study entry and upon return visits to M. D. Anderson. These samples will be used to test for certain molecules in the blood (HAMA and soluble CD20) and to check on the level of rituximab in the blood.

Treatment will be given in the hospital at the University of Texas (UT) MD Anderson. You will need to stay in the hospital for about 3 to 4 weeks. You should stay in the Houston area for about 2 to 4 weeks after the transplant. After that, you will need to return to Houston from time to time for blood tests, urine tests, and other exams.

This is an investigational study. This is an investigational study. 90Y-Zevalin is approved by the FDA for relapsed and refractory lymphoma. Its use in this trial, however, is investigational. All other drugs used in this study are FDA approved and are commercially available. Up to 60 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed CD20-positive B-cell non-Hodgkin's lymphoma (NHL) (demonstrated in lymph nodes or bone marrow), chemosensitive (at least Partial Remission (PR)).
2. No anti-cancer therapy started within three weeks, prior to study initiation, and fully recovered from all toxicities associated with prior surgery, radiation treatments, chemotherapy, or immunotherapy. No prior Rituximab within three weeks of starting therapy.
3. No prior radioimmunoconjugate therapy.
4. If patients had prior radiation, this should have not involved more than 25% of the bone marrow.
5. An IRB-approved signed informed consent.
6. Age: 18 to 65 years of age.
7. Acceptable hematologic status within two weeks prior to patient registration, including: Absolute neutrophil count ([segmented neutrophils + bands] * total white blood count (WBC)) > 1,500/mm3. Platelet counts > 100,000/mm3.
8. Patients determined to have <10% bone marrow involvement with lymphoma within four weeks before stem cell collection as defined by bilateral aspirates and biopsies.
9. Prestudy performance status of 0, 1, or 2 according to the World Health Organization (WHO).
10. Female patients included must not be pregnant or lactating.
11. Men and women or reproductive potential who are following acceptable birth control methods (as determined by the treating physician, however abstinence is not an acceptable method).
12. Patients who have previously been treated on Phase II drugs can be included if no long-term toxicity is expected, and the patient has been off the drug for four or more weeks with no significant post treatment toxicities observed
13. Patients should have at least 4 * 106 CD34+/kg peripheral stem cells collected. Whenever possible, 1 to 2 * 106 CD34+/kg, for the first 10 patients and held for 1 year in case of graft failure. If graft failure does not occur in the first 10 patients, backup cells will not be required for subsequent patients.

Exclusion Criteria:

1. Patients with impaired bone marrow reserve, as indicated by one or more of the following: Prior myeloablative therapies with autologous bone marrow transplantation (ABMT) or peripheral blood stem cell (PBSC) rescue Platelet count < 100,000 cells/mm3 Hypocellular bone marrow Marked reduction in bone marrow precursors of one or more cell lines (granulocytic, megakaryocytic, erythroid) History of failed stem cell collection of > 4*106 CD34+/kg
2. Prior radioimmunotherapy.
3. Presence of central nervous system (CNS) lymphoma.
4. Patients with chronic lymphocytic lymphoma.
5. Patients with human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS)-related lymphoma.
6. Patients with abnormal liver function: total bilirubin > 1.5 mg/dl
7. Patients with abnormal renal function: serum creatinine > 1.6 mg/dl
8. Patients who have received prior external beam radiation therapy to >25% of active bone marrow (involved field or regional).
9. Serious nonmalignant disease or infection which, in the opinion of the investigator and/or the sponsor, would compromise other protocol objectives.
10. Corrected carbon monoxide diffusion in the lung (DLCO) <50% and forced expiratory volume in 1 second (FEV1) or forced vital capacity (FVC) < 50% predicted.
11. Cardiac ejection fraction (EF) < 50% by 2-D Echogram.
12. Pleural effusions.
13. Prior radiation to lungs.
14. Abnormal cytogenetics, filter in situ hybridization (FISH) (-5, -7, 11q23)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa F. Khouri, MD,BS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chamoun K, Milton DR, Ledesma C, Young KH, Jabbour EJ, Alatrash G, Anderlini P, Bashir Q, Ciurea SO, Marin D, Molldrem JJ, Olson AL, Oran B, Popat UR, Rondon G, Champlin RE, Gulbis AM, Khouri IF. Allogeneic Transplantation after Myeloablative Rituximab/BEAM +/- Bortezomib for Patients with Relapsed/Refractory Lymphoid Malignancies: 5-Year Follow-Up Results. Biol Blood Marrow Transplant. 2019 Jul;25(7):1347-1354. doi: 10.1016/j.bbmt.2019.02.022. Epub 2019 Mar 1. PMID 30826465
- [Derived] Chahoud J, Sui D, Erwin WD, Gulbis AM, Korbling M, Zhang M, Ahmed S, Alatrash G, Anderlini P, Ciurea SO, Oran B, Fayad LE, Bassett RL Jr, Jabbour EJ, Medeiros LJ, Macapinlac HA, Young KH, Khouri IF. Updated Results of Rituximab Pre- and Post-BEAM with or without 90Yttrium Ibritumomab Tiuxetan during Autologous Transplant for Diffuse Large B-cell Lymphoma. Clin Cancer Res. 2018 May 15;24(10):2304-2311. doi: 10.1158/1078-0432.CCR-17-3561. Epub 2018 Feb 23. PMID 29476021
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 30, 2003 to September 17, 2007. All participants enrolled at the University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Y Zevalin + BEAM: Rituxan 250 mg/m2 preceding imaging dose of 111In Zevalin (5 mCi); additional infusion 250 mg/m2 Rituxan followed by therapeutic dose of 0.4 mCi/kg 90Y Zevalin received one week after Rituxan/111In Zevalin infusions. One week later, chemotherapy received with 1,3-bis(2-chloroethyl)-1-nitrosourea bis-chloronitrosourea (BCNU) (300 mg/m2, intravenously (IV) day -6) VP-16 (200 mg/m2 IV every 12 hours, days -5 to -2) cytarabine (200 mg/m2 IV every 12 hours, days -5 to -2) and melphalan (140 mg/m2 IV day -1). Autologous stem cell infused on day 0 then Rituximab 1000 mg/m2 on days +1, and +8 post transplantation.
Period: Overall Study
Arm/Group | Y Zevalin + BEAM
Started | 40
Completed | 36
Not Completed | 4
Not completed — Disease Progression | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Y Zevalin + BEAM: Rituxan 250 mg/m2 preceding imaging dose of 111In Zevalin (5 mCi); additional infusion 250 mg/m2 Rituxan followed by therapeutic dose of 0.4 mCi/kg 90Y Zevalin received one week after Rituxan/111In Zevalin infusions. One week later, chemotherapy received with BCNU (300 mg/m2, intravenously (IV) day -6) VP-16 (200 mg/m2 IV every 12 hours, days -5 to -2) cytarabine (200 mg/m2 IV every 12 hours, days -5 to -2) and melphalan (140 mg/m2 IV day -1). Autologous stem cell infused on day 0 then Rituximab 1000 mg/m2 on days +1, and +8 post transplantation.
Arm/Group | Y Zevalin + BEAM
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 53 [31 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Median
Description: Overall survival reported as number of days participants alive following treatment up to 5 years with annual follow up till disease progression. Evaluations done every 3 months for 1 year and then every 6 months for 5 years to check on the status of the disease, with long-term follow up as needed.
Time Frame: Participant followed from baseline treatment to 5 years, with study total period 8 years (study duration)
Measure: Median (Full Range); unit: days
Arm/Group | Y Zevalin + BEAM
Number analyzed (Participants) | 40
days | 1299 [8 to 2017]

2. Primary Outcome: 3-Year Overall Survival
Description: Number of participants alive 3 years following treatment. Evaluations done every 3 months for 1 year and then every 6 months to check on the status of the disease.
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Y Zevalin + BEAM
Number analyzed (Participants) | 40
percentage of participants | 78

ADVERSE EVENTS:
Time Frame: Adverse event reporting 21 days prior to autologous stem cell transplantation (ASCT) to 8 days post transplant. Overall participation period (inclusive of Y Zevalin, BEAM/Rituximab treatment and ASCT) from March 2004 to November 2011.
Arm/Group | Y Zevalin + BEAM
Serious Adverse Events (participants affected / at risk) | 7/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Y Zevalin + BEAM (N=40)
Death not related to Common Toxocity Adverse Events (CTCAE) (General disorders) | 1
Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Secondary Graft Failure (General disorders) | 1
Infection (Infections and infestations) | 2
Death due to Septic Shock (General disorders) | 1
Stem cell Infusion Reaction (Immune system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Y Zevalin + BEAM (N=40)
Alanine Aminotransferase (ALT) Increase (Metabolism and nutrition disorders) | 12
Mucositis (Gastrointestinal disorders) | 37
Diarrhea (Gastrointestinal disorders) | 29
Fever (Infections and infestations) | 3
Hypotension (Cardiac disorders) | 3
Hypertension (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 29
Vomiting (Gastrointestinal disorders) | 5
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Increased Bilirubin (Metabolism and nutrition disorders) | 6
Alkaline Phosphatase Elevated (Metabolism and nutrition disorders) | 10
Skin Rash (Skin and subcutaneous tissue disorders) | 5
Headache (Nervous system disorders) | 2
Urinary Frequency (Renal and urinary disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No